CLINICAL TRIAL: NCT04079686
Title: Single Dose Versus 24 Hours Antibiotic Prophylaxis in Reduction Mammaplasty: a Randomized Clinical Trial
Brief Title: Single Dose Versus 24 Hours Antibiotic Prophylaxis in Reduction Mammaplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Francescato Veiga (Other)
Responsible Party: Sponsor-Investigator, Daniela Francescato Veiga, Associate Professor, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PosDoc
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Plastic Surgery; Mammaplasty; Anti-bacterial Agents; Prophylaxis; Wound Infection
MeSH Terms: conditions — Wound Infection | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cephazolin (Experimental): Patients will receive antibiotics (1g cephazolin) intravenously at the anesthestic induction and every 6 hours for 24 hours
  Interventions: Drug: Cephazolin
- Sterile saline (Placebo Comparator): Patients will receive antibiotics (cephazolin) only at the anesthesia induction, and sterile saline intravenously every 6 hours for 24 hours
  Interventions: Other: Sterile saline

INTERVENTIONS:
Drug: Cephazolin — Patients undergoing reduction mammaplasty will receive 1g of cephazolin intravenously anesthetic induction and postoperatively every 6 hours, for 24 hours.
  Arms: Cephazolin
Other: Sterile saline — Patients undergoing reduction mammaplasty will receive 1g of cephazolin intravenously anesthetic induction and intravenous sterile saline postoperatively, every 6 hours, for 24 hours.
  Arms: Sterile saline

SUMMARY:
Setting: Translacional Surgery Graduation Program - Universidade Federal de São Paulo and Hospital das Clínicas Samuel Libânio - Universidade do Vale do Sapucaí. Background: Breast reduction is one of the most performed plastic surgery procedures. Antibiotics are widely prescribed, on an empirical basis, to prevent surgical site infections. However, there is a lack of evidence to support its use. Objective: To compare the influence of the use of prophylatic antibiotics as a single dose or for 24 hours on surgical site infection rates following reduction mammaplasty. Methods: Randomized trial of non-inferiority, with two parallel groups, double blinded. A total of 146 breast hypertrophy patients, with reduction mammaplasty already scheduled, will be enrolled. Patients will be randomly allocated to group A, that will receive antibiotics only at the anesthesia induction (n=73), or to group B, that will receive antibiotics at the anesthesia induction and for 24 hours (n=73). None of the patients will receive antibiotics after hospital discharge. Patients will be followed-up weekly, for 30 days, regarding surgical site infection. The Centers for Disease Control and Prevention criteria will be applied. A statistical analysis of the data will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 60 years of age
* body mass index (BMI) between 19 and 30 kg/m2
* breast hypertrophy according to the criteria of Sacchini et al. and Franco and Rebello

Exclusion Criteria:

* patients who had previously undergone another surgical procedure of the breast
* patients who have been diagnosed with a breast pathology
* smokers
* patients who had a child or breastfed within the last year
* patients with uncontrolled comorbidities, such as arterial hypertension or diabetes
* use of immunosuppressants
* patients who had any infection during the follow-up period, requiring the use of antibiotics
* patients who present any adverse effects due to the antibiotics during the study
* patients who miss follow-up assessments
* patients who withdraw their consent at any time

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2019-08-04 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with surgical site infection (SSI) | 30 days
  Patients will be monitored for the occurrence of SSI once weekly during the first 30 days following hospital discharge by a single surgeon who is blinded to their treatment group. SSI will be evaluated based on the definition adopted by the Centers for Disease Control and Prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela F Veiga, MD, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Hospital das Clinicas Samuel Libânio, Universidade do Vale do Sapucaí, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veiga DF, da Silva Garcia E, Moreira-Filho JW, de Mattos Andrade EB, Juliano Y, Veiga-Filho J, Ferreira LM. Single dose versus 24 h antibiotic prophylaxis in reduction mammaplasty: study protocol for a randomized controlled trial. Trials. 2020 Jul 2;21(1):605. doi: 10.1186/s13063-020-04539-0. PMID 32616026
- [Derived] Veiga DF, Garcia ES, Veiga-Filho J, Fialho SV, Fortunato Borges AS, Dornelas GV, Machado AA, Felix GAA, Ferreira LM. Single-Dose versus 24-Hour Antibiotic Prophylaxis in Reduction Mammaplasty: A Randomized Controlled Trial. Plast Reconstr Surg. 2025 Dec 1;156(6):835-842. doi: 10.1097/PRS.0000000000012263. Epub 2025 Aug 25. PMID 40857697
- See also: Study Protocol — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7331275/pdf/13063_2020_Article_4539.pdf